CLINICAL TRIAL: NCT00000188
Title: Selegiline in Treatment of Cocaine Dependence
Brief Title: Selegiline in Treatment of Cocaine Dependence - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, James Cornish, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-00144-2; 3R01DA012268 (NIH); K20-00144-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Dependence; Selegiline
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Selegiline

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Selegiline

SUMMARY:
The purpose of this study is to assess selegiline as a pharmacotherapy for cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1994-09; Primary Completion 1995-10 (Actual); Study Completion 1995-10 (Actual)

PRIMARY OUTCOMES:
Retention
Cocaine use
Cocaine craving

CONTACTS AND LOCATIONS:
Overall Officials: James Cornish, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- PDVAMC Treatment Research Center, Philadelphia, Pennsylvania, United States